CLINICAL TRIAL: NCT01052987
Title: A Randomized, Double-Blind, Crossover, Pharmacodynamic and Pharmacokinetic Drug Interaction Study of Tranilast in Combination With Allopurinol Compared With Tranilast Alone and Allopurinol Alone in Healthy Subjects With Hyperuricemia
Brief Title: Study of Tranilast Alone or in Combination With Allopurinol in Subjects With Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nuon Therapeutics, Inc. (Industry)
Responsible Party: Nuon Therapeutics Clinical Trials Contact, Nuon Therapeutics
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A3008GT
Record Dates: First submitted 2010-01-05; First posted 2010-01-21 (Estimated); Last update posted 2011-01-06 (Estimated); Status verified 2011-01

CONDITIONS: Gout; Hyperuricemia
Keywords: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — tranilast; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Tranilast (Experimental): Tranilast tablets
  Interventions: Drug: Tranilast
- Allopurinol (Active Comparator): Allopurinol tablets
  Interventions: Drug: Allopurinol
- Combination (Experimental): Tranilast plus Allopurinol
  Interventions: Drug: Combination - Tranilast and Allopurinol
- High dose Allopurinol (Active Comparator): 400 mg Allopurinol
  Interventions: Drug: 400 mg Allopurinol
- High dose combination (Experimental): Combination of Tranilast 300 mg and Allopurinol 400 mg
  Interventions: Drug: High dose combination

INTERVENTIONS:
Drug: Tranilast — Tranilast tablets, 300 mg, QD
  Arms: Tranilast
Drug: Allopurinol — Allopurinol tablets 300 mg, QD
  Arms: Allopurinol
Drug: Combination - Tranilast and Allopurinol — Tranilast, 300 mg QD; Allopurinol 300 mg QD
  Arms: Combination
Drug: 400 mg Allopurinol — 400 mg Allopurinol administered once daily for 7 days
  Arms: High dose Allopurinol
Drug: High dose combination — Combination of Tranilast 300 mg once daily for 7 days plus Allopurinol 400 mg once daily for 7 days
  Arms: High dose combination

SUMMARY:
This is a randomized, double-blind, 3-period 3-treatment crossover followed by a 2-period 2-treatment crossover, phase 2 study in patients with documented hyperuricemia to evaluate the effect of tranilast on allopurinol pharmacokinetics (PK) and pharmacodynamics (PD) and to evaluate the effect of allopurinol on tranilast PK and PD as measured by reduction in serum uric acid levels.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21 to 70
* Subjects with hyperuricemia who are otherwise healthy

Exclusion Criteria:

* Pregnant or nursing
* Known history of gout unless approved by the Investigator or Sponsor
* Clinically significant infection at Screening
* Known sensitivity to tranilast or allopurinol

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Mean percent decrease in serum uric acid levels | Seven days

SECONDARY OUTCOMES:
Analysis of pharmacokinetic parameters (AUC, Cmax) of tranilast, allopurinol and combination | Seven days

CONTACTS AND LOCATIONS:
Overall Officials: Director, Nuon Clinical Trials Group, Study Director — Nuon Therapeutics, Inc.
Locations (3):
- United States (3):
  - Nuon Investigative Site, Honolulu, Hawaii
  - Nuon Investigative Site, Evansville, Indiana
  - Nuon Investigative Site, Dallas, Texas